CLINICAL TRIAL: NCT01820351
Title: BICEPS FEMORIS AND VASTUS LATERALIS MUSCLE ARCHITECTURE AFTER A CHRONIC STRETCHING PROGRAM
Brief Title: Assessment of Thigh Muscle After a Stretching Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Kelly Mônica Marinho e Lima, Kelly Lima of Federal University of Rio de Janeiro, Universidade Federal do Rio de Janeiro
Purpose: Basic Science
Other Study IDs: Ethics Committee 023/11; Ethics Committee 023/11 (Other: Ethics Committee 023/11)
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Assessment of Muscle Architecture and Tendon After Chronic Stretching Program

INTERVENTIONS:
Other: static stretching exercise on 3 times a week during 8 weeks. Sets number: three of 30 seconds with intervals of equal duration

SUMMARY:
The purpose of this study is to establish, through ultrasound, measurements of the thigh muscles (Biceps Femoris and Vastus Lateralis)and the chronic effects of a static stretching program on the muscle-tendon unit these muscles.

ELIGIBILITY:
Inclusion Criteria:

* physically active male volunteers
* soldiers of the Army School of Physical Education of Rio de Janeiro, Brazil
* young men

Exclusion Criteria:

* any musculoskeletal disorder in the lower limbs
* neurological or cardiovascular disease experienced previous to or reported during the study.

Ages: 17 Years to 25 Years | Sex: Male
Age Groups: Child, Adult
Dates: Start 2011-02; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Thigh Muscle After a Stretching Program | after 8 weeks that static stretching protocol was applied

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil